CLINICAL TRIAL: NCT00371046
Title: The Use of Fetal Fibronectin and Transvaginal Ultrasound Cervical Length in Women With Threatened Preterm Labor:A Randomized Trial
Brief Title: Does Fetal Fibronectin and Ultrasound Cervical Length Help in the Evaluation of Women With Suspected Preterm Labor?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: O4U.289
Record Dates: First submitted 2006-08-31; First posted 2006-09-01 (Estimated); Last update posted 2007-03-02 (Estimated); Status verified 2007-03

CONDITIONS: Preterm Birth
Keywords: preterm labor; transvaginal ultrasound cervical length; fetal fibronectin; preterm birth
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Transvaginal ultrasound cervical length
Procedure: Cervicovaginal fetal fibronectin

SUMMARY:
The objective of this study is to investigate the effect of the use of both sonographic cervical length (CL) and fetal fibronectin (FFN) on the length of outpatient triage and preterm labor interventions in symptomatic women with intact membranes.

We performed a randomized trial of the use of transvaginal ultrasound cervical length and fetal fibronectin in women being evaluated for suspected PTL at a gestational age between 24 and 33 weeks 6 days. Women are randomized to either a standard (blinded) or a protocol arm. Women in the standard arm are evaluated without the results of the CL and FFN while women in the protocol arm are evaluated using the results of the CL and FFN and managing physicians are asked to follow a specific PTL algorithm to determine a women's eligibility for treatment. The primary outcome is length of stay in the triage area before discharge.

DETAILED DESCRIPTION:
Patients presenting with signs and symptoms suggestive of preterm labor (PTL) represent a clinical challenge. Many studies have shown that over 70% of women evaluated for PTL do not deliver within 7 days and almost 40% of women, whether they are treated or not, deliver at term. On the other hand, about 20% of women who are not thought to be in PTL will deliver preterm. Women who are diagnosed with PTL are exposed to a variety of evidenced and non-evidenced based interventions including hospital admission, tocolysis, antenatal steroids, maternal transfer and bedrest. These interventions are associated with both maternal risks and increased health care costs and often have harmful social, financial and psychological effects on the mother as well her family. Therefore, methods to accurately evaluate the risks of preterm delivery in symptomatic women would help to identify those who would most benefit from standard clinical interventions and help reduce their use in those women who would not deliver preterm. A number of retrospective and cohort studies have demonstrated that the use of fetal fibronectin (FFN) and transvaginal sonographic cervical length (TVU CL) improves prediction over standard digital exams, and that the combination of the two adds prognostic information in women admitted for PTL.

The objective of this study was to investigate the effect of the use of both sonographic cervical length and fetal fibronectin on the length of outpatient triage and preterm labor interventions in symptomatic women with intact membranes.

Methods:

Study design This is a randomized trial of the use of transvaginal ultrasound cervical length and fetal fibronectin in women being evaluated for suspected PTL on labor and delivery at the Thomas Jefferson University Hospital, Philadelphia between November 2004 and April 2006. The study was approved by the Internal Review Board.

Gestational age was assigned by last menstrual period and first or early second trimester ultrasound. If the last menstrual period was unknown or there was a discrepancy regarding the dates, the ultrasound dating was used. Eligible women who agreed to participate in the study were randomized to either a standard or a protocol arm. At the time this study was initiated neither FFN nor CL were routinely used in the management of symptomatic women presenting to L&D to be evaluated for PTL. Women in the standard arm were evaluated without the results of the CL and FFN while women in the protocol arm were evaluated using the of the CL and FFN and managing physicians were asked to follow a specific PTL algorithm to determine a women's eligibility for treatment. Physicians were encouraged to manage protocol patients according to the study recommended protocol for the use of FFN and CL, which was reviewed with them for each patient on labor and delivery by a study investigator. Once eligible for treatment, the management of PTL was then left to the discretion of the physician.

Definitions and study procedures

Before randomization all patients being evaluated for preterm labor were monitored in the triage area and uterine activity and fetal heart rate evaluated. A speculum exam was performed to rule out ruptured membranes and to obtain a specimen for fetal fibronectin. Specimens for fetal fibronectin were obtained with a Dacron swab from the posterior vaginal fornix and placed in buffer which then held on labor and delivery until the patient was either randomized, determined to be ineligible or declined to participate in the study. After randomization the specimen was immediately analyzed in our in house laboratory. Samples were delivered to the laboratory within 1 hour of obtaining the sample and results were available within 1 hour. Samples containing 50 ng or more per milliliter were designated as positive. The FFN was delayed for 24-36 hours as needed if the patient had intercourse, a pelvic exam or a transvaginal ultrasound within 24 hours. A digital exam was then performed to determine dilatation and effacement of the cervix.

Results of the fibronectin analysis were labeled by one of the study investigators after randomization so that only results from non-blinded specimens would be available to the managing physicians.

Randomization was performed by means of computer generated random blocks of numbered sealed opaque envelops which were stratified in two groups based on gestational age < 28 weeks and ≥ 28 weeks. Each envelope was opened sequentially within each strata by one of the study investigators.

Following randomization, transvaginal ultrasound assessment of the cervix was performed. Measurements were obtained using a 5-7.5 Mhz transvaginal probe placed in the anterior fornix after emptying the bladder. The transducer was oriented to obtain a sagittal view of the cervix, with the long axis view of the echogenic endocervical mucosa along the length of the canal. The probe was withdrawn slightly until the image was blurred, and enough pressure then reapplied to restore the image. CL was measured from the internal to the external os along the endocervical canal. At least three measurements were recorded over 5 minutes and the shortest best measurement in millimeters was used for the study.

Using a two-sided t-test with alpha of 0.05, we calculated that a sample size of 45 patients in each group would have an 80% power to detect a 1 hour (33%) in the mean time on labor & delivery (from 3.0 hrs to 2.0 hrs, assuming a standard deviation of 1.0). These assumptions were based on a survey taken from the Labor and Delivery triage database for the 6 months prior to the study.

ELIGIBILITY:
Inclusion Criteria:

1. gestational age between 24 and 33 weeks 6 days
2. contractions ≥ 6/hr, uterine irritability, or symptoms such as cramping, pressure, backache with or without documented contractions which prompted evaluation for PTL
3. cervical dilatation < 3cm and < 100% effacement
4. intact membranes.

Exclusion criteria:

1. ruptured membranes
2. known congenital anomaly
3. triplets or greater;
4. vaginal bleeding
5. cervical dilatation ≥ 3cm or complete effacement;
6. cerclage
7. known short cervix Women transferred on tocolytics were also excluded

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2003-10; Study Completion 2006-12

PRIMARY OUTCOMES:
Length of time for evaluation for preterm labor

SECONDARY OUTCOMES:
Admission for preterm labor
Preterm delivery less than 37 weeks
Preterm delivery less than 34 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amen Ness, MD, Principal Investigator — Thomas Jefferson University; Vincenzo Berghella, MD, Study Director — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States